CLINICAL TRIAL: NCT03199352
Title: Comparison of Hand-sewn and Linear-stapled Roux-en-Y Gastric Bypass: Outcomes in Stricture, Ulceration, and Gastritis
Brief Title: Hand-sewn and Linear-stapled Roux-en-Y Gastric Bypass: Outcomes
Status: Withdrawn | Type: Observational
Why Stopped: No participants enrolled
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0280-17-FB
Record Dates: First submitted 2017-06-22; First posted 2017-06-26 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Roux-en-y Anastomosis Site

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RYGB: Hand-sewn: This group would receive a Roux-en-y gastric bypass with the anastomosis hand-sewn using a minimally-invasive robotic surgical approach
  Interventions: Other: RYGB hand-sewn
- RYGB: linear-staple: This group would receive a Roux-en-y gastric bypass with the anastomosis sewn with a linear stapler using a laparoscopic surgical approach
  Interventions: Other: RYGB linear-staple

INTERVENTIONS:
Other: RYGB hand-sewn — Patients will have the RYGB anastomosis hand-sewn
  Groups: RYGB: Hand-sewn
Other: RYGB linear-staple — Patients will have the RYGB anastomosis performed using a linear staple.
  Groups: RYGB: linear-staple

SUMMARY:
The technique of laparoscopic Roux-en-Y gastric bypass (RYGB) has evolved significantly over the past few decades to minimize complication risks such as strictures. Three different anastomotic techniques are currently widely used hand-sewn (HS), linear-stapled (LS) and circular stapled (CS). Studies are contradictory as to the best technique to avoid complications. Many studies have focused on the stricture and infection rates of these procedures, and minimized the examination of ulceration, gastritis, and anastomotic leak. The purpose of this study is to prospectively examine how the use of linear-stapled and hand-sewn anastomotic techniques affect complication rates of marginal ulceration, gastritis, leak and stricture in patients who undergo RYGB. The goal of this study is to compare the long-term complication rates between hand-sewn robotic RYGB and linear-stapled laparoscopic RYGB. Eligible patients are men and women age 19-65 who are to undergo RYGB, have a BMI between 35-45, and RYGB is the primary procedure. The main outcomes to be measured are complications in marginal ulceration, gastritis, leak, and stricture rate at 2 and 6 weeks, and 3, 6, 9, 12, and 24 months postoperatively.

DETAILED DESCRIPTION:
1. Screening and Informed Consent Subjects will be screened on a weekly basis for eligibility of enrollment. If eligible, patients will be approached by study staff at the initial surgical consultation. The purpose of the study and risks of the procedures will be explained to the subject and the consent process must be documented accordingly in the medical record. Subjects who agree to study participation must sign an IRB approved informed consent form. Subjects will be informed that their participation in this study is voluntary and they may refuse to participate or discontinue from the study at any time. Subjects will be given the opportunity to ask the investigator questions so that they are adequately informed about the research. A copy of the signed informed consent must be provided to the subject and the informed consent process will be documented in source documents. If new information becomes available that may affect a subject's decision to continue to take part in the study, this information will be discussed with the subject by the investigator.

Failure to meet submission requirements:

Each patient will be required to meet their individual insurance companies requirements for submission of bariatric surgery approval. Subjects who provide study consent but then do not submit for insurance approval or are denied will be considered "discontinued" and will not require additional study follow-up visits. The reason for the discontinuation will be clearly delineated on the applicable case report form. Subjects in whom the robotic RYGB procedure is begun but not completed will be considered "discontinued" once discharged from the hospital and not require any additional study follow-up visits. Reasons for discontinuation will be recorded in the case report form. Additionally, female patients of child bearing age will undergo a standard of care pregnancy test at the time of the pre-operative surgical testing (2/3 weeks before surgery) and always the morning of surgery by urine HCG.

Surgical Procedures:

The operation will be performed per standard of care for both the laparoscopic RYGB and the robotic RYGB. The main difference between the two procedures is that in the robotic procedure, the intestinal anastomosis will be hand-sewn and in the laparoscopic RYGB, the anastomosis will be performed using a linear staple. Subjects will be maintained on a low-calorie diet for the first post-operative month, as per standard of care. In addition, multivitamin supplements, calcium, and iron should be prescribed and maintained per standard of care.

Schedule:

Subjects will be evaluated preoperatively, during the procedure, at discharge, and at 2 weeks, 6 weeks, 3 months, 6 months, 9 months, and 12 months. Assessments to be conducted/data collected at each visit are listed below and in the study assessments table.

1. Pre-operative Assessment

   The following assessments will be performed pre-operatively prior to the scheduled surgical procedure and the results recorded on the appropriate subject report form:

   Verification of pre-operative eligibility criteria Subject demographics (gender, age, race, ethnicity, smoking history) Height, weight, and body mass index (BMI) Comorbidity assessment (prevalence and duration of type 2 diabetes mellitus, sleep apnea, hypertension, dyslipidemia/hyperlipidemia, and other clinically relevant comorbidities as determined by the treating physician), including medications Fasting labs (glucose, hemoglobin, HbA1C, hematocrit, ferritin, albumin, total protein, calcium, parathyroid hormone, vitamin A, Vitamin B1, Vitamin B12, Vitamin D2/3, Vitamin 3, Vitamin K, folic acid, insulin, lipid panel, triglycerides, total cholesterol, high-density lipoprotein (HDL), low-density lipoprotein (LDL), C-peptides, iron, copper, and zinc) Surgical history Health- related Quality of life, as measured by the SF-36 assessment Gastrointestinal symptom rating scale, as measured by the GSRS form GERD HR-QL Pre-operative Dietary Restrictions
2. Operative Assessment The following procedures and assessments will be performed on the day of/during the procedure: Weight and BMI American Society of Anesthesiologists (ASA) grade operative time (defined as skin to skin time) anesthesia start and stop time estimated blood loss adverse events surgical technique surgical conversions to open concomitant procedures performed during the procedure
3. Discharge Assessment

   The following procedures and assessments will be performed prior to discharge:

   Length of hospital stay Surgical site infection assessment Surgical site infection (SSI) Adverse events (see below)
4. Post-operative follow-up assessments

   The following procedures and assessments will be performed at 2 weeks, 6 weeks, 3 months, 6 months, 9 months and 12 months post procedure (+/- 7 days for 2 and 6 week follow-up, +/- 14 day days for all other months).

   Post-operative standard of care:

   Compliance with prescribed dietary supplements Weight and BMI EWL Comorbidity assessment (prevalence and duration of type 2 diabetes mellitus, sleep apnea, hypertension, dyslipidemia/hyperlipidemia, and other clinically relevant comorbidities as determined by the treating physician), including medications and relevant lab tests per standard of care at 3, 6, and 12 months (glucose, hemoglobin, HbA1C, hematocrit, ferritin, albumin, total protein, calcium, parathyroid hormone, vitamin A, Vitamin B1, Vitamin B12, Vitamin D2/3, Vitamin 3, Vitamin K, folic acid, insulin, lipid panel, triglycerides, total cholesterol, high-density lipoprotein (HDL), low-density lipoprotein (LDL), C-peptides, iron, copper, and zinc) Surgical site infection assessment at 1 month only health-related quality of life (HR-QOL) (SF-36), GERD-HRQL and GSRS questionnaire expressed as change from baseline at 3, 6 and 12 months only EGD at 1 year to assess stricture, marginal ulceration, and gastritis adverse events (see below)
5. Adverse Events Adverse events for all bariatric procedures are tracked within our centers Metabolic and Bariatric Surgery Accreditation and Quality Improvement Program (MBSAQIP) database. All bariatric centers accredited by the American Society for Metabolic and Bariatric Surgery (ASMBS) are required to submit all bariatric surgery data to the MBSAQIP database for quality review. Our bariatric surgery team has open access to our centers data for quality review purposes and will compare adverse events for the robotic and laparoscopic RYGB to the other procedures performed by our center. Adverse events are categorized by organ system (wound, respiratory, urinary tract, CNS, cardiac, or other) as specified by the MBSAQIP. Any post-operative occurrence within 30 days will be documented if related to the bariatric procedure. Bariatric related readmission and reoperations are also tracked per MBSAQIP guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 19-70 who will receive their weight loss procedure at UNMC
* BMI of 35-45
* RYGB as the primary procedure

Exclusion Criteria:

* RYGB performed as a revisional procedure
* Prior foregut surgery
* H/o smoking, unless the patient quit more than 10 years ago
* Complication of bariatric procedure post-operatively that would significantly affect weight loss (extended period of TPN, clinically significant leak, major organ failure, severe protein malnutrition or failure to thrive)

Ages: 19 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Eligible participants who have access to care at UNMC.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2020-11-12 (Actual)

PRIMARY OUTCOMES:
Stricture Rate | 1 year
  Examine the development of stricture at the anastomosis. Stricture will be determined by esophagogastroduodenoscopy (EGD) at 1 year post-surgery.

SECONDARY OUTCOMES:
Leak rate | 1 year
  Examine leak development at the anastomosis site. Leak is determined by clinical findings of pain, tachycardia, fever, and confirmed by a barium swallow study that indicates a hole at the anastomosis site
Quality of Life impact | 1 year
  Examine the quality of life impact of the surgery, using the SF-36 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Vishal Kothari, MD, Principal Investigator — University of Nebraska

IPD SHARING:
Plan to Share IPD: No
We do not currently plan to make individual participant data available to other researchers.